CLINICAL TRIAL: NCT04056975
Title: A Phase I, Single Centre, Open-label, Dose-escalation Study of A-319 in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: Study of A-319 in Patients With Relapsed or Refractory B-cell Lymphoma
Acronym: A-319
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EVIVE Biotechnology (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP071744
Record Dates: First submitted 2019-07-08; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): A-319 dosage: 0.05, 0.15, 0.03, 0.06, 0.12, 0.18, 0.24 μg/kg
  Interventions: Biological: Recombinant Anti-CD19m-CD3 Antibody Injection

INTERVENTIONS:
Biological: Recombinant Anti-CD19m-CD3 Antibody Injection — Intravenous Infusion

SUMMARY:
Title: A Phase I, Single Centre, Open-label, Dose-escalation Study of A-319 in Patients With Relapsed or Refractory B-cell Lymphoma

DETAILED DESCRIPTION:
Protocol Number: SP071744 Study Stage: Phase I Study Number: 1 site Subject Number: up to 54 patients with Relapsed or Refractory B-cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, all genders
* Patients with definite B-cell Lymphoma, includes FL, MZL, MCL, DLBCL.
* Patients With Relapsed or Refractory B-cell Lymphoma
* ECOG ≤ 2
* Lesions are measurable in 21 days before treatment
* Normal bone marrow function
* Normal liver, kidney, lung and heart function
* the Subjects can sign the ICF and obey the protocol, elsewise, his/her guardian should sign
* Life expectancy is at least 3 months

Exclusion Criteria:• Past or present CNS disease

* Associated with lymphoma by the infiltrates of CNS
* A history of autoimmune disease with CNS involvement or autoimmune disease
* Previous history of autoimmune disease or other malignancy
* A history of deep venous thrombosis or pulmonary embolism
* Auto-HSCT was performed within 12 weeks prior to initiation of treatment
* Previous organ transplantation or allogeneic hematopoietic stem cell transplantation
* The Investigator determined that the patients were associated with a disease, medical condition, or social factor that might affect study results or compliance
* Immunosuppressant are being used
* Radiotherapy was given within 6 weeks prior to A-319 treatment
* Chemotherapy, immunotherapy and targeted therapy were received within 4 weeks before A-319 treatment
* Previous CAR-T cell therapy
* Received anti-lymphoma drugs in the first 4 weeks of A-319 treatment
* There was no recovery of toxic effects (CTCAE> grade 1 adverse events) at the last treatment, except hair loss
* Those who underwent major surgery 28 days before enrollment (excluding lymph node biopsy);Or plan to operate during the study period
* Those who had received active/attenuated live vaccine within 28 days prior to screening
* For pregnant (positive pregnancy test) and lactating women, those of childbearing age who signed the informed consent form and did not agree to use contraception for at least 3 months after the end of the study;Within 7 days prior to the first day of treatment, women of childbearing age require a positive serum pregnancy test (HCG)
* Male patients who signed informed consent forms and did not agree to use contraception for at least 3 months at the end of the study (except surgical sterilization)
* Known allergy to immunoglobulin or research drugs and their excipients
* Patients considered unfit to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-27 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Incidence and Characteristics of SAE of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle 1 (each cycle is 28 days)
  Incidence and Characteristics of SAE
Evaluate the MTD and DLT of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle 1 (each cycle is 28 days)
  dose limited toxicity(DLT), maximum tolerance dose(MTD)

SECONDARY OUTCOMES:
Evaluate the PK(Cmax) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  Peak Plasma Concentration(Cmax)
Evaluate the PK(AUC) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  Area under the plasma concentration versus time curve(AUC)
Evaluate the PK(Tmax) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  time to peak (Tmax)
Evaluate the PK(T1/2) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  half-life time(T1/2)
Evaluate the PK(CL) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  clearance(CL)
Evaluate the PK(Vz) of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  volume of distribution(Vz)
Evaluate the PD of A-319 Treat on Relapsed or Refractory B-cell Lymphoma | At the end of Cycle3 (each cycle is 28 days)
  B-cell level

CONTACTS AND LOCATIONS:
Overall Officials: Song Yuqin, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Yes
all IPD
Supporting Information: SAP, CSR
Time Frame: After 20January2022(estimated), for 1years(estimated).
Access Criteria: All.